CLINICAL TRIAL: NCT05987553
Title: The Influence of an E-learning Program on Recognition of Actinic Keratosis by General Practitioners). Implementation of Actinic Keratosis Guidelines Among General Practitioners.
Brief Title: The Influence of an E-learning Program on Recognition of Actinic Keratosis
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1334
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Actinic Keratoses; E-learning; Dermatology
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General practitioners: All participants were general practitioners (in training).
  Interventions: Other: e-learning program

INTERVENTIONS:
Other: e-learning program — All participants participate in this intervention: an e-learning program about the recognition of actinic keratosis. The program exists of 30 cases. Each case exists of a question and thorough explanation including references to various sources.

SUMMARY:
The evaluation on the diagnostic accuracy of actinic keratosis recognition by general practitioners before and after participation on an e-learning program.

DETAILED DESCRIPTION:
Actinic keratosis is defined as the most frequent common intra-epithelial neoplasm in the Caucasian population, with an increasing prevalence. If left untreated, actinic keratosis has the potency to develop into a cutaneous squamous-cell carcinoma. Treatment of actinic keratosis is aimed at both lesion reduction and to prevent malignant transformation. To achieve treatment adherence for patients, it is necessary to raise physician awareness about actinic keratosis.

This study primarily aimed to investigate whether the sensitivity of establishing a correct actinic keratosis diagnosis by general practitioners (in training) would increase after participating in an e-learning program about the recognition of actinic keratosis. This was achieved by comparing the results of a pre- and post-test completed by general practitioners which was incorporated in the e-learning program.

ELIGIBILITY:
Inclusion Criteria:

* general practitioner in the Netherlands
* access to e-learning module via phone/computer/tablet
* knowledge of the Dutch language

Exclusion Criteria:

* no knowledge of the Dutch language
* different specialists than general practitioner

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from general practitioners who
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in sensitivity | Measurement by baseline and after finalising the e-learning program (same day up until 30 days)
  Difference in sensitivity of participants in the recognition of actinic keratosis, before and after the use of an e-learning program (paired).
Difference in specificity | Measurement by baseline and after finalising the e-learning program (same day up until 30 days)
  Difference in specificity of participants in the recognition of actinic keratosis, before and after the use of an e-learning program (paired).

SECONDARY OUTCOMES:
Difference in area under the receiver operating characteristic (ROC) curve | Measurement by baseline and after finalising the e-learning program (same day up until 30 days)
  Difference in area under the curve of participants in the recognition of actinic keratosis, before and after the use of an e-learning program.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, prof.dr., Principal Investigator — Maastricht UMC
Locations (1):
- Ellen Oyen, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No